CLINICAL TRIAL: NCT05091398
Title: Erector Spinae Plane, Paravertebral Versus Intercostal Nerve Block for VATS Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Mogahed, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 34779/7/21
Record Dates: First submitted 2021-10-01; First posted 2021-10-25 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Thoracic
Keywords: Erector spinae plane; paravertebral; intercostal nerve block; VATS

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): ultrasound-guided erector spinae block on T4 and T6 levels after the anesthesia induction and turning the patient in the lateral position
  Interventions: Other: Regional analgesia of thoracic surgical patients
- Group II (Active Comparator): ultrasound-guided paravertebral block on T4 and T6 levels after the anesthesia induction and turning the patient in the lateral position
  Interventions: Other: Regional analgesia of thoracic surgical patients
- Group III (Active Comparator): ultrasound-guided intercostal nerve block on T4 and T6 levels after the anesthesia induction and turning the patient in the lateral position
  Interventions: Other: Regional analgesia of thoracic surgical patients

INTERVENTIONS:
Other: Regional analgesia of thoracic surgical patients — ultrasound-guided erector spinae block on T4 and T6 levels ,paravertebral block or intercostal nerve block after the anesthesia induction and turning the patient in the lateral position with 30 mL 0.5% bupivacaine +50 µ adrenaline will be injected by the surgeon through the thoracoscope .

SUMMARY:
The optimal analgesia method in video-assisted thoracoscopic surgery (VATS) remains controversial. 105 patients scheduled to undergo video-assisted thoracic surgery under general anesthesia will be included. Patients will be randomly allocated to receive ultrasound-guided ESP blocks on T4 and T6 levels (Group ESPB, n = 35),PVB (Group PVB, n = 35) after the anesthesia induction and turning the patient in the lateral position or (Group ICNB, n=35) with 30 mL 0.5% bupivacaine +50 µ adrenaline will be injected by the surgeon through the thoracoscope .

DETAILED DESCRIPTION:
Standard general anesthesia was applied Patients will be randomly allocated to receive single shot of ESP blocks (Group ESPB), Paravertebral blocks (Group PVB) or (Group ICNB )at T4 and T6 levels according to a random number list that will be generated by a computer and will be stored in sealed envelopes. An independent experienced anesthesiologist will perform the first two blocks or surgeon will perform the third one through the thoracoscope according to the random number. The study coordinator, attending anesthesiologist, data collection resident and the patients will be all blinded to the treatment group assignment. All blocks will be applied on patient's back in a lateral position. Postoperative analgesia regimen consisted of a continuous infusion of iv iboprofen and morphine as a second rescue drug. Demographic data, past medical history, surgical and anesthetic data will be documented. Postoperative pain scores, consumption of analgesia and quality of recovery will be recorded to evaluate the analgesic effect.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients
* Thoracic surgery

Exclusion Criteria:

* Coagulation defect

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
end tidal sevoflurane | 150 minutes
  intraoperative end tidal sevoflurane

SECONDARY OUTCOMES:
Blood pressure | 150 minutes
  Intraoperative blood pressure in mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Mona Mohamed Mogahed, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided